CLINICAL TRIAL: NCT02497963
Title: Foreskin Graft Tubularized Incised Plate Urethroplasty (TIP) vs Tubularized Incised Plate (TIP) for Primary Hypospadias. Randomized Clinical Trial (FGTIP-TIP)
Brief Title: Foreskin Graft Tubularized Incised Plate Urethroplasty vs Tubularized Incised Plate for Primary Hypospadias (FGTIP-TIP)
Acronym: FGTIP-TIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Byron Pacheco Mendoza, MD, MsC, Pediatric Urologist,, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIM 2015-079
Record Dates: First submitted 2015-06-25; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Foreskin Graft-Tubularized Incised Plate (Experimental): Group of patients with primary hypospadias undergoing Foreskin Graft Tubularized Incised Plate Urethroplasty. The surgery involves making an incision on the midline of the urethral plate, graft inner foreskin, and create a new urethra on a urethral catheter.
  Interventions: Procedure: Foreskin Graft-Tubularized Incised Plate
- Tubularized Incised Plate (Active Comparator): Group of patients with primary hypospadias undergoing Tubularized Incised Plate Urethroplasty. The surgery involves making an incision on the midline of the urethral plate, and create a new urethra on a urethral catheter.
  Interventions: Procedure: Tubularized Incised Plate

INTERVENTIONS:
Procedure: Foreskin Graft-Tubularized Incised Plate — TIP Urethroplasty with foreskin graft in primary hypospadias
  Arms: Foreskin Graft-Tubularized Incised Plate
Procedure: Tubularized Incised Plate — TIP Urethroplasty without foreskin graft in primary hypospadias
  Arms: Tubularized Incised Plate

SUMMARY:
The purpose of this study is to determine the efficacy and safety of tubularized incised plate urethroplasty versus foreskin graft tubularized incised plate urethroplasty in primary hypospadias. This study only included patients with width of urethral plate ≤ 7 mm, width of glans ≤ 14 mm, and urethral plate depth shallow o moderate.

DETAILED DESCRIPTION:
Urethroplasty technique more used in the world for hypospadias repair is Tubularized Incised Plate described by Snodgrass in 1994. Kolon and Gonzales described a technical modification to the TIP in 2000, which is called grafting foreskin.

There are characteristics of the glans and urethral plate favoring the development of complications. In this study the researchers include patients with primary hypospadias, with these characteristics above, and compare two surgical techniques: TIP vs FG-TIP.

The main aim is to determine the efficacy (functional and cosmetic) and safety (complications) of TIP vs FG-TIP.

The study design is a randomized clinical trial, double blind (patient and evaluator), parallel groups.

The sample size was calculated comparing two proportions, with a alpha 0.05, beta 0.2; 34 patients per group. The main outcome is complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hypospadias without previous surgery
* Hypospadias with width of urethral plate ≤ 7 mm, width of glans ≤ 14 mm, and urethral plate depth shallow o moderate.

Exclusion Criteria:

* Patients diagnosed with hypospadias and severe psychomotor development delay
* Patients with disorders of sexual development without gender assignment

Ages: 3 Months to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with complications as a measure of safety | Fourth month after surgery

SECONDARY OUTCOMES:
Proportion of participants with fistula as a measure of safety | Fourth month after surgery
Proportion of participants with stricture as a measure of safety | Fourth month after surgery
Proportion of participants with breakdown as a measure of safety | Fourth month after surgery

OTHER OUTCOMES:
Degree of Cosmetic by HOPE Score as a measure of efficacy | Fourth and sixth months after suregry
Urinary mean flow by uroflowmeter as a measure of efficacy | Fourth and sixth months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mario E Rendón Macías, MD MsC, Study Chair — CMNXXI, IMSS; Onofre Muñoz Hernández, MD MsC, Study Director — Hospital Infantil de Mexico Federico Gomez

REFERENCES:
- [Background] Snodgrass WT. Re: Effect of suturing technique and urethral plate characteristics on complication rate following hypospadias repair: a prospective randomized study O. Sarhan, M. Saad, T. Helmy and A. Hafez J Urol 2009; 182: 682-686. J Urol. 2010 Apr;183(4):1649-50; discussion 1650. doi: 10.1016/j.juro.2009.12.048. Epub 2010 Mar 4. No abstract available. PMID 20206364
- [Result] Snodgrass W. Tubularized, incised plate urethroplasty for distal hypospadias. J Urol. 1994 Feb;151(2):464-5. doi: 10.1016/s0022-5347(17)34991-1. PMID 8283561
- [Result] Kolon TF, Gonzales ET Jr. The dorsal inlay graft for hypospadias repair. J Urol. 2000 Jun;163(6):1941-3. PMID 10799234
- [Result] Holland AJ, Smith GH. Effect of the depth and width of the urethral plate on tubularized incised plate urethroplasty. J Urol. 2000 Aug;164(2):489-91. PMID 10893631
- [Result] Mouravas V, Filippopoulos A, Sfoungaris D. Urethral plate grafting improves the results of tubularized incised plate urethroplasty in primary hypospadias. J Pediatr Urol. 2014 Jun;10(3):463-8. doi: 10.1016/j.jpurol.2013.11.012. Epub 2013 Dec 10. PMID 24360521